CLINICAL TRIAL: NCT00011687
Title: US Study of Semen Quality in Partners of Pregnant Women
Brief Title: Study for Future Families
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9916-CP-001
Record Dates: First submitted 2001-02-26; First posted 2001-02-28 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Pregnancy
Keywords: Fertility; Hormones; Semen; Reproductive Health

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The Study for Future Families is a multi-center study that is recruiting pregnant women and their partners in four US cities to look for differences between cities in several measures of reproductive health. These measures include how long it took couples to conceive as well as hormone levels and semen quality in the male partners. This study is modeled after a study in four European cities so that,when complete, data on the 300 couples in each of the eight cities can be compared.

ELIGIBILITY:
Pregnant women and their partners who are literate in English or Spanish and competent to complete a questionnaire whose pregnancy was conceived without medical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400
Dates: Start 1999-09; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States